CLINICAL TRIAL: NCT06809010
Title: grouP O wholE blooD (LTO-WB): storagE leSion impacT And infLammation
Brief Title: grouP O wholE blooD : storagE leSion impacT And infLammation
Acronym: PEDESTAL EFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Collaborators: Centre de transfusion sanguine des Armées, Clamart, France (Unknown); INSERM, SAINBIOSE U1059 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 241-PEDESTAL EFS; 2024-A01405-42 (Other: ANSM (Agence Nationale de Sécurité du Médicament et des produits de santé))
Record Dates: First submitted 2025-01-08; First posted 2025-02-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Blood Donation; Blood Platelets; Blood Donors; Inflammation; Transfusion
Keywords: blood; LTO-WB; characterization of labile blood products; whole blood; apheresis; plasma; platelet; red blood cells; inflammation; transfusion
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: The first 15 participants will be whole blood donations and the next 15 apheresis donations. Working sequentially on whole blood donations (n=15) followed by apheresis donations (n=15) will enable us to evaluate the biological markers of interest on whole blood donations and not repeat these experiments on apheresis platelet donations, which are rarer and longer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole blood (Other): Participants in this arm donate whole blood
  Interventions: Biological: Whole blood donation
- Apheresis (Other): Participants in this arm make a plasma/platelet apheresis donation
  Interventions: Biological: Apheresis donation

INTERVENTIONS:
Biological: Whole blood donation — This intervention involves the collection of a whole blood bag.
  Arms: Whole blood
Biological: Apheresis donation — This procedure involves the collection of a plasma/platelets bag by apheresis
  Arms: Apheresis

SUMMARY:
"Etablissement Français du Sang" (EFS) prepares labile blood products from blood donations that are separated by type (red blood cells, plasma and platelets).

The "Centre de Transfusion Sanguine des Armées" (CTSA) produces an innovative labile blood product, LTO-WB, corresponding to group O leukocyte-free whole blood.

The objective of the PEDESTAL EFS study is to compare the inflammatory and biological characteristics of blood products prepared by the EFS vs. the labile blood product prepared by the CTSA.

DETAILED DESCRIPTION:
Hemorrhage is one of the main causes of preventable death among soldiers in combat. Currently, the majority of patients receive blood components (red blood cells, platelets, plasma) rather than whole blood. These factors lead doctors deployed on external operations (OPEX) to use plasma, RBCs and platelets. However, platelet concentrates may not be available on missions, as their storage conditions and shelf life are not always compatible with OPEX logistics. The only solutions to this problem is to use group O leucocyte-depleted whole blood without hemolysin (or Low Titer O Whole Blood, LTOWB), which provides the three elements in physiological proportions. However, while studies have shown this product to be effective in stopping bleeding, its inflammatory potential, linked to the presence of platelets, has not yet been investigated. Indeed, in addition to their hemostatic role, platelets are also involved in inflammation.

The main objective of our research project is to deploy in vitro and in vivo tools to compare LTOWB, focusing on its inflammatory component with conventional and well-mastered transfusion products for (1) platelet-related inflammation (LTOWB vs. Buffy coat pooled platelet concentrate or single donor apheresis platelet concentrates), (2) RBC-related inflammation (LTOWB vs. RBC concentrates) and (3) other circulating inflammatory molecules (LTOWB vs. fresh frozen plasma).

The definition of biomarkers is essential to optimize the use of these products, depending on the therapeutic indication. Linking these biomarkers with the effectiveness of transfusions will help to determine the risk/benefit ratio of transfusions that may be required in rural and austere environments, such as OPEX in comparison to civilian transfusion medicine.

ELIGIBILITY:
Inclusion Criteria:

Self-referred donors eligible for blood donation (whole blood and/or platelet/plasma apheresis), meeting the following inclusion criteria:

* Be in good health
* Weigh at least 50 kg
* Must be between 18 and 70 years of age for whole blood donation and between 18 and 65 years of age for plasma/platelet donation by apheresis.

Exclusion Criteria:

Subjects ineligible to donate blood

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the platelet-related inflammatory potential of blood products throughout storage. | Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 14, Day 21, Day 28, Day 35 and Day 42
  Assessment of the platelet-related inflammatory potential throughout storage, including the concentration of platelet-related soluble immunomodulatory molecules and the cellular expression of activation markers, which characterize the quality of labile blood products, notably apheresis platelet concentrates, standard Buffy coat pooled platelet concentrate, red blood cell concentrates and fresh plasma prepared by EFS, compared to platelet, red blood cells and plasmas from LTO-WB.
  Several techniques will be used to this purpose, including ELISA, Luminex multi-analyte profiling for soluble immunomodulatory molecule assessment and flow cytometry for activation marker cellular expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Maison du don de l'EFS Auvergne Rhônes-Alpes, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: SAINBIOSE INSERM U1059 - SAnté INgéniérie BIOlogie St-Etienne — https://sainbiose-lab.fr/